## **Cover Page for Statistical Analysis Plan**

Official Title: Rural Tailored COVID-19 Communication and SARS-CoV-2 Antibody

Testing Evaluation and Uptake

NCT Number: NCT06085547

Date: December 12, 2024

## **Statistical Analysis Plan:**

The primary analysis for all self report study outcomes is based on assessing mean differences across the two study arms. Our arms include rural residents who are assigned either to the general (group 1) or rural targeted (group 2) antibody video group. A series of independent samples t-tests were conducted for all interval level/self-report outcomes, which included Theory of Planned Behavior and rural-adapted anticipatory racism measures. We also computed Cohen's d effect sizes to consider practical significance of pairwise differences. Subsequent analyses will explore sociodemographic variables and individual differences, such as gender and rural identity, as potential moderators of group differences. Future exploratory considerations will utilize hierarchical moderated multiple regression procedures.

For dichotomous (yes-no) outcomes related to accepting and completing the antibody test kit we conducted two group chi square goodness of fit tests.

Please feel free to contact me at <a href="mailto:lucastod@msu.edu">lucastod@msu.edu</a> with any questions.

Thank you,

Todd Lucas, PhD
C.S. Mott Endowed Professor of Public Health
Charles Stewart Mott Department of Public Health
College of Human Medicine, Michigan State University